CLINICAL TRIAL: NCT07192354
Title: The Relationship Between Cyberchondria and Health Perception and Anxiety Level in Pregnant Women: A Cross-sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Nurcan Contarli, Lecturer, Karabuk University
Other Study IDs: KBUPTherapy
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cyberchondria; Pregnancy
MeSH Terms: interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Participants will be administered the Cyberchondria Severity Scale Short Form (CSS-12), Health Perception Scale, and State and Trait Anxiety Scale online via Google form.

SUMMARY:
Pregnancy is a unique period in which women require extensive health information both to protect their own health and to prepare for motherhood. The literature indicates that pregnant women most frequently seek information on healthy nutrition, physical activity, fetal development, pregnancy symptoms, childbirth preparation, vaccination, and medication use. Although health professionals are considered reliable sources of information, due to limited accessibility, pregnant women often turn to the internet and social media. This increases the risk of exposure to inaccurate or incomplete information and may sometimes lead to cyberchondria. Moreover, during pregnancy, factors such as educational level, socioeconomic conditions, and family relationships contribute to the frequent occurrence of anxiety disorders, which can negatively affect the mother's quality of life and fetal development. Health perception, on the other hand, is an important concept that shapes individuals' health behaviors and responsibilities. However, studies examining the relationship between cyberchondria, anxiety levels, and health perception in pregnant women are limited. This study aims to reveal the relationship between health information-seeking behaviors, health perception, and anxiety levels in this special population of pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older, pregnant, have access to the internet at any time, and have the ability to use it.
* Must be proficient in Turkish to understand the scales.

Exclusion Criteria:

* Having a diagnosed psychiatric illness,
* Being a healthcare worker,
* Having cognitive impairment or mental or physical limitations to the extent that they cannot understand questions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10-27 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
The Cyberchondria Severity Scale | 1 month
  The Cyberchondria Severity Scale (CSS) was originally developed by McElroy and Shevlin (2014) to evaluate cyberchondria, defined as a form of anxiety characterized by excessive health-related information seeking on the internet. Subsequently, McElroy et al. (2019) introduced the short form of the scale, the CSS-12. The Turkish adaptation, validity, and reliability study of the CSS-12 was conducted by Söyler et al. (2021).
  The CSS-12 consists of 12 items, each rated on a 5-point Likert-type scale ranging from 1 ("never") to 5 ("always"). Total scores are calculated by summing all item responses, with possible scores ranging from 12 to 60. Higher scores indicate greater severity of cyberchondria. The scale does not contain any reverse-coded items. The CSS-12 comprises four subdimensions: excessiveness, distress, reassurance-seeking, and compulsion.
The Health Perception Scale | 1 month
  The Health Perception Scale (HPS) was developed by Diamond et al. in 2007 to assess individuals' perceptions of their own health. The Turkish adaptation, including validity and reliability testing, was conducted by Kadıoğlu et al. in 2012. The scale consists of 15 items rated on a 5-point Likert-type scale, with response options ranging from "Strongly Disagree" to "Strongly Agree." Negative items are reverse-coded (Strongly Disagree = 5 to Strongly Agree = 1). The scale includes four subdimensions: central control, self-awareness, certainty, and importance of health. Total scores range from 15 to 75, with higher scores reflecting a more positive health perception. Participants indicate their agreement with each item, allowing researchers to quantify their overall health perception and examine its relationship with other psychosocial variables.
State-Trait Anxiety Inventory | 1 month
  The State-Trait Anxiety Inventory (STAI) was originally adapted into Turkish by Öner and Le Compte between 1974 and 1977 to evaluate anxiety levels in both adolescent and adult Turkish populations. The inventory is widely used in research involving young and adult groups. The State Anxiety Scale items assess the intensity of feelings or behaviors in response to specific situations, with responses rated on a 4-point scale: 1 = Not at all, 2 = Somewhat, 3 = Much, 4 = Completely. The Trait Anxiety Scale items evaluate the frequency of feelings or behaviors over time, with response options: 1 = Almost never, 2 = Sometimes, 3 = Often, 4 = Almost always. The State Anxiety Scale consists of both direct items (3, 4, 6, 7, 9, 12, 13, 14, 17, 18) and reverse-scored items (1, 2, 5, 8, 10, 11, 15, 16, 19, 20). Similarly, the Trait Anxiety Scale includes direct items (22, 23, 24, 25, 28, 29, 31, 32, 34, 35, 37, 38, 40) and reverse-scored items (21, 26, 27, 30,

CONTACTS AND LOCATIONS:
Overall Officials: Tarik OZMEN, PhD, Study Chair — Karabuk University; Nesibe Sumeyye KUTAHYALIOGLU, PhD, Principal Investigator — Karabuk University; Nurcan CONTARLI, PhD, Principal Investigator — Karabuk University
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No